CLINICAL TRIAL: NCT05659303
Title: Evaluation of an Outpatient Protocol in Patients Operated for Laparoscopic Hysterectomy
Acronym: HYSTECOE
Status: Completed | Type: Observational
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Responsible Party: Sponsor
Other Study IDs: GCS RAMSAY SANTE
Record Dates: First submitted 2022-12-13; First posted 2022-12-21 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Hysterectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Laparoscopic hysterectomy: Patient having undergone a hysterectomy, planned as an outpatient during the pre-operative consultation, by laparoscopic route.
  Interventions: Procedure: Laparoscopic hysterectomy

INTERVENTIONS:
Procedure: Laparoscopic hysterectomy — Patient having undergone a hysterectomy, planned as an outpatient during the pre-operative consultation, by laparoscopic route.

SUMMARY:
Removal of the uterus, or hysterectomy, is a surgical operation that involves partial or total removal of the uterus. It can be done by vaginally, laparoscopically or laparotomically.

Since the first hysterectomy performed by laparoscopy in 1989, this approach has gained popularity to varying degrees depending on the countries. This technique allows a major surgical procedure to be performed by incisions of only a few millimeters, thus reducing parietal pain and visceral in addition to a cosmetic benefit.

Since 2013, more than 200 laparoscopic hysterectomies have been scheduled on an outpatient basis at the Clinique des Cèdres (France). The analysis of this retrospective series of approximately 200 patients would provide elements related to the practice of laparoscopic hysterectomy in ambulatory in France.

DETAILED DESCRIPTION:
Removal of the uterus, or hysterectomy, is a surgical operation that involves partial or total removal of the uterus. It can be done by vaginally, laparoscopically or laparotomically.

Since the first hysterectomy performed by laparoscopy in 1989 (Reich, 1989), this approach has gained popularity to varying degrees depending on the countries. This technique allows a major surgical procedure to be performed by incisions of only a few millimeters, thus reducing parietal pain and visceral in addition to a cosmetic benefit. Thus, when we offer women requiring a two-way hysterectomy first, 84% of them prefer the laparoscopic route to the laparotomy route (Nieboer, 2009). Alongside this surgical advance, an improvement in anesthesy techniques combined with the use of anti-inflammatories and antiemetics made it possible to improve the speed of recovery and therefore the possibility of a departure early, but not premature, from the hospital. In the United States, a study published in 2012 (Schiavone, 2012) reported the hospital stays of more than 128,000 women who underwent a laparoscopic total hysterectomy and reported that 46% of them had been operated on as an outpatient.

Since 2013, more than 200 laparoscopic hysterectomies have been scheduled on an outpatient basis at the Clinique des Cèdres.

The analysis of this retrospective series of approximately 200 patients would provide elements related to the practice of laparoscopic hysterectomy in ambulatory in France.

ELIGIBILITY:
Inclusion Criteria:

* Female aged 18 or over.
* Patient having undergone a hysterectomy, planned as an outpatient during the pre-operative consultation, by laparoscopic route with or without adnexectomy, for benign or malignant reasons, at the Clinique des Cèdres since 2013.
* Patient having been informed of the research and not objecting to the use of his data as part of this research

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Study Population: Female aged 18 or over having undergone a hysterectomy, planned as an outpatient during the pre-operative consultation, by laparoscopic route with or without adnexectomy, for benign or malignant reasons, at the Clinique des Cèdres since 2013.
Sampling Method: Non-Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2022-10-15 (Actual); Primary Completion 2023-07-17 (Actual); Study Completion 2023-07-17 (Actual)

PRIMARY OUTCOMES:
Rate of performance, on an outpatient basis, of the laparoscopic hysterectomy procedure | 1 day
  Success rate of performance, on an outpatient basis, of the laparoscopic hysterectomy procedure, on all laparoscopic hysterectomies scheduled on an outpatient basis since 2013 at the Clinique des Cèdres

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique des Cèdres, Cornebarrieu, France

IPD SHARING:
Plan to Share IPD: No